CLINICAL TRIAL: NCT05522270
Title: Concentrated Growth Factor Versus Platelet Rich Fibrin in Revitalization of Necrotic Young Permanent Incisors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmad Elheeny (Other)
Responsible Party: Sponsor-Investigator, Ahmad Elheeny, clinical professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 320
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: double (participant,outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- revitalization by concentrated growth factor (Experimental): modified platelet concentrate
  Interventions: Procedure: revitalization by concentrated growth factor
- revitalization by platelet rich fibrin (Active Comparator): platelet concentrate
  Interventions: Procedure: revitalization by concentrated growth factor

INTERVENTIONS:
Procedure: revitalization by concentrated growth factor — modified platelet concentrate
  Other Names: revitalization by platelet rich fibrin

SUMMARY:
Regenerative endodontic procedures (REPs) are the most recent proposal to manage immature permanent teeth with necrotic pulps. So in this study, the investigator will evaluate the clinical and radiographical revitalization success in necrotic young permanent anterior teeth of participants by using Concentrated Growth Factor versus Platelet-Rich Fibrin

DETAILED DESCRIPTION:
has been entered

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with immature permanent incisors
* Presence of clinical signs and symptoms of necrosis or chronic apical periodontitis. The chronic apical periodontitis signs and symptoms include little discomfort with intermittent episodes of pus discharge through the sinus tract.

Exclusion Criteria

1. Abnormal tooth mobility.

* Positive history of allergic reaction, systemic diseases, severe emotional or behavioral problems.
* Unrestorable teeth
* Abnormal tooth mobility
* Children with systemic, severe behavioral, or emotional problems

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | one year
  Regaining tooth vitality with electric pulp testing Clinical examination includes pain absence, normal tooth mobility, and no sensitivity to percussion
Radiographic success using Periapical index (PAI) | one year
  Criteria of PAI scores:
  score "1" normal periapical structure score "2" small changes in bone structures score "3" changes in bone structure with some mineral loss score "4" periodontitis with well-defined radiolucent area score "5" severe periodontitis with exacerbating features

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months